CLINICAL TRIAL: NCT04521309
Title: Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2) Antibodies Based Intravenous Immunoglobulin (IVIG) Therapy for Severe and Critically Ill COVID-19 Patients
Brief Title: SARS-CoV-2 Antibodies Based IVIG Therapy for COVID-19 Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Higher Education Commission (Pakistan) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: biotech001
Record Dates: First submitted 2020-05-07; First posted 2020-08-20 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: COVID19 ( Corona Virus Disease -2019); SARS-CoV-2 (Severe Acute respiratory syndrome Coronavirus 2); Passive Immunization; Intravenous Immunoglobulin (IVIG); Pooled convalescent Plasma; Critically ill COVID-19 patients; Severe COVID-19 patients; Antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Standard care only n = 10 patients.
- IVIG dose: 0.15 g/kg (Experimental): Standard Care + Single dose of 0.20 g/Kg anti-COVID-19 IVIG (experimental drug prepared at DUHS) n= 10 patients
  Interventions: Biological: SARS-CoV-2 antibody based IVIG therapy
- IVIG dose: 0.20 g/kg (Experimental): Standard Care + Single dose of 0.25 g/Kg anti-COVID19 IVIG (experimental drug prepared at DUHS) n= 10 patients
  Interventions: Biological: SARS-CoV-2 antibody based IVIG therapy
- IVIG dose: 0.25 g/kg (Experimental): Standard Care + Single dose of 0.30 g/Kg anti-COVID19 IVIG (experimental drug prepared at DUHS) n= 10 patients
  Interventions: Biological: SARS-CoV-2 antibody based IVIG therapy
- IVIG dose: 0.30 g/kg (Experimental): Standard Care + Single dose of 0.35 g/Kg anti-COVID19 IVIG (experimental drug prepared at DUHS) n= 10 patients
  Interventions: Biological: SARS-CoV-2 antibody based IVIG therapy

INTERVENTIONS:
Biological: SARS-CoV-2 antibody based IVIG therapy — Patient groups will receive IVIG prepared from pooled convalescent plasma from recovered COVID-19 patients. This will be administered sequentially and in varying dosages, infused over a period of 12 hours, intravenously.Additionally, all treatment groups will receive same standard care as control group. Standard Care as per hospital protocol, which may include:
  Airway support, Anti-Viral medication, Antibiotics, Fluid Resuscitation, Hemodynamic Support, Steroids, Painkillers, Anti-Pyretics
  Arms: IVIG dose: 0.15 g/kg; IVIG dose: 0.20 g/kg; IVIG dose: 0.25 g/kg; IVIG dose: 0.30 g/kg

SUMMARY:
Severe and critically ill patients will be enrolled in the study (50 patients) after duly filled consent forms. Recipients shall be divided in to 5 groups with 10 patients per group to compare clinical efficacy and safety of patients in clinical phase I/phase II study. Each group shall receive particular single dose of Intravenously administered Immunoglobulins (IVIG) developed from convalescent plasma of recovered COVID-19 individual , an experimental drug along with standard treatment except for control group which will receive standard treatment only.

DETAILED DESCRIPTION:
Passive immunization using intravenous immunoglobulins (IVIG) has been tested for treating previous viral outbreaks and holds the potential to save lives in the current crisis. Recently researchers from China reported satisfactory recovery of critically ill Corona Virus Disease 2019 (COVID 19) patients when high dose intravenous immunoglobulin (IVIG) were administered.

Research team at Dow University of Health Sciences has purified immunoglobulin (both SARS-CoV 2 antibodies and existing antibodies) from convalescent plasma of COVID19 individuals and pooled to prepared IVIG formulation to treat severe and critically ill COVID-19 patients. To evaluate safety of the formulation animal (rats) safety trials and survival of all the animals were observed.

It is intended to assess safety and efficacy of experimental the IVIG treatment in severe and critically ill COVID 19 patients through phase I/phase II randomized single blinded clinical trial with fifty study participants. FDA outlined criteria for passive immunization using convalescent plasma, which will be used for recruiting participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Have positive SARS-CoV-2 PCR on nasopharyngeal and/or oropharyngeal swabs
* Admitted in isolation ward and ICU of institutes affiliated with DUHS
* have severe or critical COVID 19 as judged by the treating physician
* Consent given by the patient or first degree relative

Exclusion Criteria:

* Pregnancy
* Previous allergic reaction to immunoglobulin treatment
* Ig A deficiency
* Patient requiring 2 inotropic agents to maintain blood pressures
* Known case of any autoimmune disorder
* Acute kidney injury or chronic renal failure
* Known case of thromboembolic disorder
* Aseptic meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
28 Days mortality | 28 days
  All cause mortality of participants will be monitored for 28 days to assess the safety and efficacy of IVIG treatment.
Requirement of supplemental oxygen support | 28 days
  Number of days required for invasive or non-invasive oxygen supply during hospital stay as per oxygen saturation status of patient
Number of days on assisted ventilation | 28 days
  Number of days a participant will be requiring assisted ventilation both invasive and noninvasive
Days to step down | 28 days
  Shifting from ICU to ward
Days to Hospital Discharge | 28 days
  Duration from day of enrollment in study to Day of hospital discharge
Adverse events during hospital stay | 28 days
  Kidney failure, hypersensitivity with cutaneous or hemodynamic manifestations, aseptic meningitis, hemolytic anemia, leuko-neutropenia, transfusion related acute lung injury (TRALI)
Change in C-Reactive Protein (CRP) levels | 28 days
  Change in C-Reactive Protein (CRP) levels from baseline will be used to monitor inflammation
Change in neutrophil lymphocyte ratio | 28 days
  change in neutrophil lymphocyte ratio from baseline will be used to monitor inflammation

SECONDARY OUTCOMES:
Change in Ferritin levels | 28 days
  change in Ferritin level from baseline will be used to monitor inflammation and immune dysregulation
Change in lactate dehydrogenase (LDH) levels | 28 days
  change in LDH from baseline will be used to monitor infections and tissue health
Change in radiological (X-ray) findings | 28 days
  Any change seen in radiological chest X-ray findings
Days to negative SARS-CoV-2 Polymerase Chain Reaction (PCR) test | 28 days
  Time taken for participant to receive negative COVID-19 PCR test
Anti-SARS-CoV-2 Antibody | 28 days
  Anti-SARS-CoV-2 antibody titre from blood measured by semi-qualitative method
Change in fever | 28 days
  Change in body temperature from baseline will be used to monitor safety and efficacy
Change in Sodium levels | 28 days
  Change in electrolytes (Sodium) seen in participants
Change in Potassium levels | 28 days
  Change in electrolytes (Potassium) seen in participants
Change in Chloride levels | 28 days
  Change in electrolytes (Chloride) seen in participants
Change in Bicarbonate levels | 28 days
  Change in electrolytes (Bicarbonate) seen in participants

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Shaukat Ali, PhD, Principal Investigator — Dow University of Health Sciences, Principal Dow College of Biotechnology
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham AC, Goh HP, Koh D. Treatment of COVID-19: old tricks for new challenges. Crit Care. 2020 Mar 16;24(1):91. doi: 10.1186/s13054-020-2818-6. No abstract available. PMID 32178711
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Buchacher A, Iberer G. Purification of intravenous immunoglobulin G from human plasma--aspects of yield and virus safety. Biotechnol J. 2006 Feb;1(2):148-63. doi: 10.1002/biot.200500037. PMID 16892245
- [Background] Hughes RA, Donofrio P, Bril V, Dalakas MC, Deng C, Hanna K, Hartung HP, Latov N, Merkies IS, van Doorn PA; ICE Study Group. Intravenous immune globulin (10% caprylate-chromatography purified) for the treatment of chronic inflammatory demyelinating polyradiculoneuropathy (ICE study): a randomised placebo-controlled trial. Lancet Neurol. 2008 Feb;7(2):136-44. doi: 10.1016/S1474-4422(07)70329-0. PMID 18178525
- [Background] Hung IFN, To KKW, Lee CK, Lee KL, Yan WW, Chan K, Chan WM, Ngai CW, Law KI, Chow FL, Liu R, Lai KY, Lau CCY, Liu SH, Chan KH, Lin CK, Yuen KY. Hyperimmune IV immunoglobulin treatment: a multicenter double-blind randomized controlled trial for patients with severe 2009 influenza A(H1N1) infection. Chest. 2013 Aug;144(2):464-473. doi: 10.1378/chest.12-2907. PMID 23450336
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Pandey S, Vyas GN. Adverse effects of plasma transfusion. Transfusion. 2012 May;52 Suppl 1(Suppl 1):65S-79S. doi: 10.1111/j.1537-2995.2012.03663.x. PMID 22578374
- [Derived] Ali S, Uddin SM, Shalim E, Sayeed MA, Anjum F, Saleem F, Muhaymin SM, Ali A, Ali MR, Ahmed I, Mushtaq T, Khan S, Shahab F, Luxmi S, Kumar S, Arain H, Khan M, Khan AS, Mehmood H, Rasheed A, Jahangeer A, Baig S, Quraishy S. Hyperimmune anti-COVID-19 IVIG (C-IVIG) treatment in severe and critical COVID-19 patients: A phase I/II randomized control trial. EClinicalMedicine. 2021 Jun;36:100926. doi: 10.1016/j.eclinm.2021.100926. Epub 2021 Jun 4. PMID 34109306
- [Derived] Ali S, Uddin SM, Ali A, Anjum F, Ali R, Shalim E, Khan M, Ahmed I, M Muhaymin S, Bukhari U, Luxmi S, Khan AS, Quraishy S. Production of hyperimmune anti-SARS-CoV-2 intravenous immunoglobulin from pooled COVID-19 convalescent plasma. Immunotherapy. 2021 Apr;13(5):397-407. doi: 10.2217/imt-2020-0263. Epub 2021 Feb 9. PMID 33557591
- [Derived] Ali S, Luxmi S, Anjum F, Muhaymin SM, Uddin SM, Ali A, Ali MR, Tauheed S, Khan M, Bajwa M, Baig SU, Shalim E, Ahmed I, Khan AS, Quraishy S. Hyperimmune anti-COVID-19 IVIG (C-IVIG) Therapy for Passive Immunization of Severe and Critically Ill COVID-19 Patients: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 2;21(1):905. doi: 10.1186/s13063-020-04839-5. PMID 33138867
- See also: World Health Organization (WHO) technical guidance on COVID-19 — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance
- See also: WHO guidelines for Use of Convalescent Whole Blood or Plasma Collected from Patients Recovered from Ebola Virus Disease for Transfusion, as an Empirical Treatment during Outbreaks — http://www.euro.who.int/__data/assets/pdf_file/0011/268787/Use-of-Convalescent-Whole-Blood-or-Plasma-Collected-from-Patients-Recovered-from-Ebola-Virus-Disease-for-Transfusion,-as-an-Empirical-Treatment-during-Outbreaks-Eng.pdf

DOCUMENTS (1):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT04521309/Prot_001.pdf